CLINICAL TRIAL: NCT01173146
Title: Imaging of Residual Prostate Cancer During Prostatectomy Using ProstaFluor®, a Prostate-Specific Membrane Antigen (PSMA)-Targeted Fluorescent Agent FDA Trial
Brief Title: Imaging of Residual Tumor During Prostatectomy
Status: Withdrawn | Type: Observational
Why Stopped: Costs for antibody production rose; supplemental funding request not approved.
Sponsor: Spectros Corporation (Industry)
Collaborators: Vanderbilt University (Other); Cornell University (Other)
Responsible Party: Principal Investigator, David Benaron, CEO, Spectros Corporation
Other Study IDs: PCA-002
Record Dates: First submitted 2010-07-27; First posted 2010-07-30 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Prostate Cancer
Keywords: Primary prostate cancer undergoing prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Prostate Cancer is the most common cancer in men, affecting about as many men as women diagnosed with breast cancer, and killing about as many men per year as breast cancer kills women.

The most common surgical treatment is prostatectomy, the removal of the prostate. During prostate surgery, tumor remains at the edge of the surgery, called residual tumor, in 30% of all prostatectomies. Such patients have a significantly higher risk of local recurrence of the cancer, and higher rates of death. In contrast, even patients with cancer outside of the prostate, but still nearby the prostate, do better when the margins are made clean of tumor during surgery.

The investigators propose to reduce the number of patients with residual tumor after surgery. The investigators will test in patients a fluorescent molecule that allows cancer to be detected during surgery. If this trial works as designed, the investigators will reduce the number of patients who have to receive additional treatment, such as high doses of radiation to the lower abdomen, because the amount of residual tumor left behind has been minimized. This may also lead to higher rates of survival.

This type of detection of cancer the investigators employ is called Molecular imaging. The investigators believe that molecular imaging will be the key to improved diagnosis, individualized treatment selection, and treatment monitoring.

If successful, a large human trial will be conducted after this study with a corporate imaging partner.

DETAILED DESCRIPTION:
In this 5 year academic-industrial partnership to FDA approval, an experienced team and partners including Cornell, Vanderbilt, Intuitive Surgical, LI-COR, and Sand Hill Institute, will move a prostate-targeted fluorescent contrast agent, demonstrated in animals in a prior project to allow real-time detection of residual tumor, through FDA approval to human use. The unmet need is that because prostate tumor at the surgical margin is undetectable in real time, residual tumor at the margin occurs in 30% of all prostatectomies. Such patients have a significantly higher risk of local recurrence, metastasis, and death, and also require radiation therapy. In contrast, even patients with extra-prostatic extension of tumors do better when the margins are made clean of tumor during surgery.

We propose to leverage our experience and our animal-proven agent to synthesize, receive FDA IND approval on, and Phase I/II test our targeted fluorescent conjugate in a pilot study in 96 human subjects. Our agent is made from a commercial LI-COR fluorescent dye, and a humanized antibody from Cornell and Millennium Pharmaceuticals (huJ-591). The targeted antibody tags Prostate-Specific Membrane Antigen (PSMA) which is present on the outside of all prostate cells of luminal (prostate duct) origin, and was demonstrated in prior funding to produce 4-12 fold contrast for prostate cells over nearby tissues in animals. The device will be tested a sites using a fluorescence-sensitive surgery system from Intuitive Surgical, a $10 billion robotic surgery company.

The PI of this grant has previously developed and commercialized fundamental optical technologies -- he (1) co-developed the first in vivo luciferase imaging system at Stanford and co-founded Xenogen, and (2) he developed T-Stat®, the first FDA-approved detection system for insufficient blood flow to tissue. Other team members have synthesized dye conjugates for commercial use, and managed antibody-based drug formulation through FDA approval.

The corporate partners, LiCor (a world-leader in automated sequencing instruments and reagents using near infrared devices and dyes) and Sand Hill Institute (experienced at antibody formulation), and Intuitive Surgical, provide proven commercial translational experience in contrast agents and FDA approval. These groups will formulate and synthesize the agent, leading to FDA IND filing and human clinical testing. Alternative paths minimize risks at each stage.

If successful, the commercial dye will be readied for Phase III multi-center trial with a major surgical tool partner, a costly and required path to market introduction. Major imaging companies (Siemens, Phillips, GE, and others) also have molecular imaging programs, into which this contract agent will fit. A successful imaging agent would likely be adopted. Extensions to ovarian cancer using the folate type II receptor, and other targets, are envisioned, including use with other targeting antibodies developed by other groups. We anticipate that this will be among the first of many real-time surgery-targeting optical contrast agents in human subjects. Areas with immediate application are the detection of lymphatic spread intraoperatively for prostate cancer, as well as for ovarian cancer using a Folate. We expect that the market for such a device in cancer could reasonably be in the hundreds of millions of dollars/year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Prostate Cancer
* Plan for Prostatectomy
* Signed informed consent

Exclusion Criteria:

* Informed consent not obtained

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects undergoing prostatectomy for prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of ProstaFluor® measured by Margin positivity after surgery (Phase II) | 2 weeks after surgery for each patient
  Is residual disease present in subject after surgery?
Safety of Prostafluor® (Phase I) | 6 weeks after surgery for each patient
  Testing for adverse reactions to Prostafluor

SECONDARY OUTCOMES:
Binding of ProstaFluor® to Prostate Cells as Measured in Pathology Laboratory After Prostatectomy | 96 hours after surgery
  Prostates removed will be studied during dose escalation for evidence of binding to prostate cells of luminal origin.

CONTACTS AND LOCATIONS:
Overall Officials: David Benaron, MD, Principal Investigator — Spectros Corporation
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
Study withdrawn, no data collected.